CLINICAL TRIAL: NCT04030754
Title: Comparison of Effectiveness of Amniotic Membrane and Duoderm Dressings in Pediatric Burn Patients: a Randomized Controlled Trial
Brief Title: Comparison of Effectiveness of Amniotic Membrane and Duoderm Dressings in Pediatric Burns
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fatima Numeri, Assistant Professor, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 257/RC/KEMU
Record Dates: First submitted 2019-02-26; First posted 2019-07-24 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Burns
Keywords: pediatric burns, dressings, amniotic membrane, duoderm
MeSH Terms: conditions — Burns | interventions — Biological Dressings

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amniotic membrane group (Experimental): amniotic dressing will be applied to these patients
  Interventions: Combination Product: amniotic membrane
- duoderm group (Experimental): duoderm dressing will be applied to these patients as intervention
  Interventions: Combination Product: duoderm dressing

INTERVENTIONS:
Combination Product: amniotic membrane — amniotic membrane is a biological dressing
  Arms: amniotic membrane group
Combination Product: duoderm dressing — duoderm dressing is a synthetic dressing
  Arms: duoderm group

SUMMARY:
There is a difference in frequency of wound infection, mean pain score, mean of time for skin grafting and hospital stay in pediatric 2nd and 3rd degree burns, between amniotic membrane and duoderm dressings

DETAILED DESCRIPTION:
After informed consent of the patients, patients who will fulfill the inclusion and exclusion criteria will be enrolled in the study from Department of Pediatric Surgery, Mayo Hospital Lahore and will be randomly allocated by lottery method into 2 groups by the doctor. Group A and B with 86 patients in each group. Group A patients will be undergoing amniotic membrane dressing, while group B patients will undergo colloid gel foam dressing. Basic demographic information will be noted. Effect modifiers (hemoglobin level, weight and height) will be noted.

In group A, the wounds will be washed with normal saline and then covered with amniotic membrane over which a layer of Vaseline gauze will be applied and dressing with gauze and the crape bandage will be applied. Every 3-4 days these dressings will be changed and assessed for pain, wound infection and wound c/s will be sent. Placentas from clean vaginal deliveries and elective C-sections will be taken. Blood of mother will be screened. Amniotic membrane will be separated from placenta in a clean sterile bowl. Bowl will be put in refrigerator at 4 degrees.

In group B, wound will be washed with normal saline . The wound site will be covered with Colloid Gel Foam and gauze, and crape bandage will be applied. Dressing will be changed after 3-4 days. The outcome (pain score, wound infection,time for skin grafting and hospital stay) will be compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* 10-45 % percent 2nd and 3rd degree fresh burns age less than 12 years patients of both gender

Exclusion Criteria:

* patients whose parents are not willing patients whose wound c/s comes positive at the time of admission patients who have associated medical disorder and trauma.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
mean time for skin grafting | average time will be 21 days
  time for grafting when wound has healthy granulation tissue
frequency of wound infection | at 5th day of dressing
  redness around burnt wound, tenderness, swelling, increased temperature (>4 degrees), exudation and growth on wound cultures
mean of hospital stay | at the time of discharge, that can be from 7th day to 30th day
  time at which patient wound is completely healed and no wound infection present, average time will be up to 30 days
mean of pain for patients of age <8 years assessed by Visual Analogue Score | at 5th day of dressing change
  pain will be assessed at the time of dressing change. for patients<8 years of age visual analogue score will be used.
mean of pain for patients of age >8 years assessed by Face, Leg, Activity, Cry, Consolabilty Pain Scale. | at 5th day of dressing change
  FLACC (face,leg, activity, cry, consolability) pain scale will be used

CONTACTS AND LOCATIONS:
Overall Officials: fatima naumeri, mbbs, fcps, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Ibran E, Mirza FH, Memon AA, Farooq MZ, Hassan M. Mortality associated with burn injury - a cross sectional study from Karachi, Pakistan. BMC Res Notes. 2013 Dec 19;6:545. doi: 10.1186/1756-0500-6-545. PMID 24354896
- [Background] Mohammadi AA, Johari HG, Eskandari S. Effect of amniotic membrane on graft take in extremity burns. Burns. 2013 Sep;39(6):1137-41. doi: 10.1016/j.burns.2013.01.017. Epub 2013 Mar 21. PMID 23523222
- [Background] Martin FT, O'Sullivan JB, Regan PJ, McCann J, Kelly JL. Hydrocolloid dressing in pediatric burns may decrease operative intervention rates. J Pediatr Surg. 2010 Mar;45(3):600-5. doi: 10.1016/j.jpedsurg.2009.09.037. PMID 20223327
- [Background] Eskandarlou M, Azimi M, Rabiee S, Seif Rabiee MA. The Healing Effect of Amniotic Membrane in Burn Patients. World J Plast Surg. 2016 Jan;5(1):39-44. PMID 27308239
- See also: about method of preparation and application of amniotic membrane — https://www.ncbi.nlm.nih.gov/pubmed/?term=Eskandarlou+M%2C+Azimi+M%2C+Rabiee+S+and+Rabiee+MA